CLINICAL TRIAL: NCT06726850
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Phase II Clinical Study to Evaluate the Efficacy and Safety of GS1-144 Tablets in the Treatment of Moderate to Severe Vasomotor Symptoms in Chinese Postmenopausal Women.
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of GS1-144 Tablets in the Treatment of Moderate to Severe Vasomotor Symptoms in Chinese Postmenopausal Women.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GenSci074-201
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2024-12

CONDITIONS: Vasomotor Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): Participants will receive multiple doses of placebo matching GS1-144 tablet for 12 consecutive weeks.
  Interventions: Drug: Placebo
- GS1-144 tablet (Experimental): Participants will receive multiple doses of GS1-144 tablets for 12 consecutive weeks.
  Interventions: Drug: GS1-144

INTERVENTIONS:
Drug: Placebo — In the placebo arm, participants will consume a placebo matching GenSci1-144 for 12 consecutive weeks.
  Other Names: Placebo tablet
  Arms: placebo
Drug: GS1-144 — In the GS1-144 arm, participants will receive multiple doses of GS1-144 tablets for 12 consecutive weeks
  Arms: GS1-144 tablet

SUMMARY:
A Randomized, Double-blind, Placebo-controlled, Parallel-group Phase II Clinical Study to Evaluate the Efficacy and Safety of GS1-144 Tablets in the Treatment of Moderate to Severe Vasomotor Symptoms in Chinese Postmenopausal Women.

DETAILED DESCRIPTION:
A Randomized, Double-blind, Placebo-controlled, Parallel-group Phase II Clinical Study to Evaluate the Efficacy and Safety of GS1-144 Tablets in the Treatment of Moderate to Severe Vasomotor Symptoms in Chinese Postmenopausal Women.

ELIGIBILITY:
Inclusion Criteria

* BMI is 18.5 to 30 kg/㎡(inclusive);
* Females meeting 1 of the following criteria of menopause at screening visit: spontaneous amenorrhea for ≥ 12 consecutive months, spontaneous amenorrhea for ≥ 6 consecutive months with serum follicle-stimulating hormone (FSH) > 40 IU/L, or 6 weeks past a postsurgical bilateral oophorectomy with or without hysterectomy;
* Participants who are seeking treatment or relief for VMS and meet the criteria for moderate to severe VMS symptoms: during the 7 consecutive days prior to randomization, participants must have a minimum average of 7 episodes of moderate to severe VMS symptoms per day;
* For females with uterus: endometrial thickness ≤ 4mm as shown by TVU at screening, or > 4mm without atypical hyperplasia or carcinogenesis of the endometrium from the subsequent biopsy results (If the biopsy sample is insufficient or can't be obtained, it is considered normal and meets this inclusion criterion);
* Volunteered to sign ICF and be able to understand and comply with the requirements of this study.

Exclusion Criteria:

* Diseases or dysfunctions known to interfere with the clinical trial, including but not limited to: neuropsychiatric, cardiovascular, urological, digestive, respiratory,musculoskeletal, metabolic, endocrine, haematological, immune, dermatological and oncological conditions, etc., or poorly controlled chronic diseases with clinical significance;
* Thyroid or parathyroid-related hormones abnormalites with clinical significance at screening or baseline;
* Confirmed moderate to severe liver fatty at screening or baseline;
* Any surgical or medical conditions that may significantly affect the absorption, distribution, metabolism, and/or excretion of the drug, such as a history of gastrointestinal surgery (gastrectomy, gastroenterostomy, enterectomy, etc.), urinary tract obstruction, or dysuria;
* Current or prior history of malignancy (except for malignancies and basal cell carcinoma that have not received any antineoplastic treatment within 5 years prior to screening visit, or have currently recovered or have no risk of relapse during this study as assessed by the investigator);
* Abnormal uterine bleeding with clinical significance during screening period or baseline period;
* Participants who have attempted suicide within the last 1 year or are currently at risk of impulsive behavior or suicide;
* Participants with a history of severe allergy to investigational products or any of their excipients or with allergic constitution (e.g., being allergic to two or more drugs or foods);
* Participants who have positive serology results of hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab) or syphilis;Abnormalities in vital signs during the screening period or baseline period, e.g., resting pulse rate < 55/min or > 105/min; systolic blood pressure < 90 mmHg or ≥ 160 mmHg; diastolic blood pressure < 60 mmHg or ≥ 100 mmHg, that upon evaluation by the investigator may interfere with this clinical study;
* BI-RADS (Breast Imaging Reporting and Data System) Category ≥4 on breast ultrasound within 6 months prior to randomization;
* Participants who have positive pregnancy test during screening or baseline period.
* 12-lead electrocardiography (ECG) abnormalities during screening period or baseline period, e.g., heart rate-corrected QT interval QTcF absolute value >470 ms (Fridericia's formula: QTcF=QT/RR0.33) that upon evaluation by the investigator may interfere with this clinical study;
* Abnormalities in laboratory tests during screening period or baseline period, e.g., alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2×upper limit of normal (ULN), or total bilirubin (TBIL) >1.5×ULN, that upon evaluation by the investigator may interfere with this clinical study;
* Creatinine >1.5×ULN or estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 based on modification of diet in renal disease (MDRD) during screening period or baseline period;
* The participant has used or is using prohibited medications/therapies (moderate or strong CYP1A2 inhibitors, hormone replacement therapy or any VMS therapeutic agents [prescription, non-prescription or herbal medicines]) at screening and is unwilling to discontinue and wash out such medications throughout the study (see Section 6.9 for the washout intervals for prohibited concomitant medications and prior medications);
* Having participated in any other clinical trial within 3 months or any clinical study of fezolinetant or other treatments for VMS (except for participants who have not received any investigational product) within 1 year prior to screening, or planning to participate in any other clinical trial;
* Current or prior history of drug use, drug abuse or alcohol abuse;
* Any other conditions that are unsuitable for participating in this study in the opinion of the investigator.

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in the frequency of moderate to severe VMS at Week 4. | Week 4
  VMS symptom electronic log. Patient's overall impression of change scale(PGI-C). A scale of a patient's overall impression of severity(PGI-S).Perimenopausal specific Quality of Life scale(MENQOL). Modified Kupperman scale.
Changes from baseline in the frequency of moderate to severe VMS at Week 12 | Week 12
  VMS symptom electronic log. Patient's overall impression of change scale(PGI-C). A scale of a patient's overall impression of severity(PGI-S).Perimenopausal specific Quality of Life scale(MENQOL). Modified Kupperman scale.

SECONDARY OUTCOMES:
Changes from baseline in the severity of moderate to severe VMS at Week 4 | Week 4
  VMS symptom electronic log. Patient's overall impression of change scale(PGI-C). A scale of a patient's overall impression of severity(PGI-S).Perimenopausal specific Quality of Life scale(MENQOL). Modified Kupperman scale.
Changes from baseline in the severity of moderate to severe VMS at Week 12 | Week 12
  VMS symptom electronic log. Patient's overall impression of change scale(PGI-C). A scale of a patient's overall impression of severity(PGI-S).Perimenopausal specific Quality of Life scale(MENQOL). Modified Kupperman scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided